CLINICAL TRIAL: NCT01918592
Title: PET/MRI and Biomarkers in Clinical Staging of Bladder Cancer and in the Estimation of Neoadjuvant Chemotherapy Response Prior to Radical Cystectomy
Brief Title: PET/MRI and Biomarkers in Bladder Cancer
Acronym: ACEBIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Peter Boström, chief, department of urology, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACEBIB
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; neoadjuvant chemotherapy; radical cystectomy; lymphadenectomy; biomarker
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI/PET (Experimental)
  Interventions: Device: MRI/acetate-PET imaging

INTERVENTIONS:
Device: MRI/acetate-PET imaging
  Other Names: Philips Ingenuity PET/MR device; 11C-acetate as PET-tracer

SUMMARY:
Muscle invasive bladder cancer is an aggressive malignancy. Currently the investigators lack accurate imaging technologies in clinical staging and estimation of response to neoadjuvant chemotherapy as well as prognostic biomarkers.

In the current study novel imaging modality (MRI/PET) is utilized to stage bladder cancer prior to transurethral resection of bladder-tumor and after neoadjuvant chemotherapy. Also prognostic biomarkers are studied from TUR-BT tissues, blood and urine to estimate response to neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* invasive or locally advanced bladder cancer based on cystoscopic evaluation
* Age: 18 to 85 years old
* Language spoken: Finnish or Swedish
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethical Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* Prior medical history: Patient must have no history of serious cardiovascular, liver or kidney disease
* Infections: Patient must not have an uncontrolled serious infection
* Contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* Patient refusing radical cystectomy or chemotherapy
* Intravesical Bacillus Calmette-Guerin instillations within 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
staging accuracy of PET/MRI in bladder cancer | 3 months
  Accuracy of PET/MRI to stage newly diagnosed bladder cancer. MRI/PET staging results is compared to pathology report of TUR-BT and cystectomy specimens.

SECONDARY OUTCOMES:
Accuracy of PET/MRI to estimate response to neoadjuvant chemotherapy | 3 mo
  Accuracy of PET/MRI to estimate response to neoadjuvant chemotherapy prior to radical cystectomy. MRI/PET results is compared to pathology report of cystectomy specimen.

OTHER OUTCOMES:
Accuracy of prognostic biomarkers to estimate response to neoadjuvant chemotherapy. | 6 mo
  Accuracy of tissue, blood and urine based biomarkers to estimate response to neoadjuvant chemotherapy is estimated

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Salminen A, Jambor I, Merisaari H, Ettala O, Virtanen J, Koskinen I, Veskimae E, Sairanen J, Taimen P, Kemppainen J, Minn H, Bostrom PJ. 11C-acetate PET/MRI in bladder cancer staging and treatment response evaluation to neoadjuvant chemotherapy: a prospective multicenter study (ACEBIB trial). Cancer Imaging. 2018 Aug 2;18(1):25. doi: 10.1186/s40644-018-0158-4. PMID 30068379